CLINICAL TRIAL: NCT04602663
Title: Optimal Time for Follow up After Variceal Band Ligation in Cirrhotic Patients: a Randomized Trial
Brief Title: Optimal Time for Follow up After Variceal Band Ligation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VARICES
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Esophageal Varices
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- follow up every week (Experimental): Variceal Band ligation every week.
  Interventions: Device: Esophageal Variceal Band ligation
- follow up every 2 weeks (Experimental): Variceal Band ligation every 2 weeks
  Interventions: Device: Esophageal Variceal Band ligation
- follow up every 3 weeks (Experimental): Variceal Band ligation every 3 weeks
  Interventions: Device: Esophageal Variceal Band ligation
- follow up every 4 weeks (Experimental): Variceal Band ligation every 4 weeks
  Interventions: Device: Esophageal Variceal Band ligation

INTERVENTIONS:
Device: Esophageal Variceal Band ligation — Band ligation of OV
  Other Names: Band ligation

SUMMARY:
Optimal time for follow up after variceal band ligation in cirrhotic patients remains to be determined

DETAILED DESCRIPTION:
Optimal time for follow up after variceal band ligation in cirrhotic patients remains to be determined. So, we designed this trial to answer this question.

ELIGIBILITY:
Inclusion Criteria:

* cirrhotic portal hypertension with medium or large sized or risky varices or variceal bleeding

Exclusion Criteria:

* non-cirrhotic portal hypertension

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients with eradicated varices | 1 year
  The total number of patients with eradicated varices

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Alboraie, MD, Principal Investigator — Al-Azhar University; Ahmed Maher, MD, Principal Investigator — Cairo University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No